CLINICAL TRIAL: NCT06001346
Title: ActiveCBT for Depression: Transforming Treatment Through Exercise Priming
Brief Title: CBT+ for Depression
Acronym: CBT+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jacob Meyer, Assistant Professor, Kinesiology, University of Wisconsin, Madison
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R61MH129407 (NIH); 1R61MH129407-01A1 (NIH)
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder
Keywords: Exercise Priming; Depression; Cognitive Behavioral Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ActiveCBT (Experimental): Participants will complete a standardized 30-minute exercise session on a stationary bike prior to therapy. Participants will view one of 8 standardized 30-minute nature documentary videos while exercising.
  Interventions: Behavioral: ActiveCBT
- CalmCBT (Active Comparator): Participants will view one of 8 standardized 30-minute nature documentary videos while resting quietly prior to therapy.
  Interventions: Behavioral: CalmCBT

INTERVENTIONS:
Behavioral: ActiveCBT — Participants will complete a standardized 30-minute aerobic exercise session on a stationary bicycle prior to therapy. Supervised exercise sessions will consist of steady-state exercise at a moderate intensity corresponding to a '13' or 'somewhat hard' rating of perceived exertion. Continuous monitoring of heart rate, resistance/load, and RPE will occur throughout exercise. To closely match the groups, participants will also view 30-minute nature videos while exercising.
  Arms: ActiveCBT
Behavioral: CalmCBT — Participants will view one of 8 standardized 30-minute nature videos while resting quietly prior to therapy. These are emotionally neutral videos and will allow for participants in both groups to have the same amount of attention and contact time.
  Arms: CalmCBT

SUMMARY:
This study investigates the effects of a novel intervention approach, intentionally sequencing aerobic exercise immediately prior to therapy sessions (i.e., cognitive behavioral therapy [CBT]) to determine its effects on both specific and common factors underlying the antidepressant effect of CBT (i.e., mechanisms of CBT). To assess the utility of this treatment augmentation, investigators plan to conduct a randomized controlled trial involving 40 adults with Major Depressive Disorder who will watch a nature documentary while either resting quietly (termed 'CalmCBT') or exercising at a moderate intensity ('ActiveCBT') immediately prior to 8 weekly sessions of CBT. It is hypothesized that target CBT mechanisms of antidepressant action (i.e., self-reported working alliance and behavioral activation) will be more effectively engaged by ActiveCBT vs. CalmCBT.

DETAILED DESCRIPTION:
Frontline treatments for major depressive disorder (MDD), including cognitive behavioral therapy (CBT), have limited effectiveness, with half of patients not responding to CBT and half relapsing within 2 years. Strategies that increase the potency of MDD treatments are needed. We are testing a novel treatment strategy using aerobic exercise to prime a subsequent CBT session ('ActiveCBT'). Exercise priming is hypothesized to lead to greater engagement of CBT mechanisms of action through both common and specific factors linked to depression outcomes; this CBT augmentation approach has yet to be empirically tested. The study will consist of an 8-week randomized controlled trial in 40 adults with MDD performing 30-minutes of moderate exercise or quiet rest (CalmCBT vs. ActiveCBT) prior to weekly CBT sessions. Using a time- and attention-matched control, all participants will view a standardized documentary series for these 30 pre-therapy minutes with the only difference between groups being exercise or calmly resting. This project will also employ machine learning and natural language processing via the Lyssn platform to objectively evaluate the language and words used during therapy. The overall goals are to: 1) demonstrate exercise priming effects on target CBT mechanisms, 2) link psychological and neuroplastic exercise priming to CBT mechanisms, and 3) explore the sensitivity of objective machine learning-based markers from Lyssn to ActiveCBT-induced therapy differences. This trial will establish the potential for a subsequent confirmatory efficacy trial to rigorously test the potential of exercise priming to enhance treatment. If this innovative, biologically-informed approach successfully 'primes' subsequent therapy, this could be used to augment other treatments and in other disorders, significantly improving mental health treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with DSM-5 MDD, confirmed via SCID.
* Having current depressive symptoms of at least mild severity defined by HAM-D rating ≥8.
* Being between age 18 and 65.
* Either not engaging in any mental health treatment (e.g., medication, psychological, or behavioral) OR on a stable mental health treatment regimen and willing to maintain it for the length of the intervention.
* Willing and safe to exercise based on the Physical Activity Readiness Questionnaire.
* Being CBT-naïve (as defined by never undergoing structured CBT).

Exclusion Criteria:

* currently pregnant, nursing, or planning to become pregnant,
* severe obesity (BMI=40)
* diagnosed with lifetime or current Psychosis, Mania, or Bipolar Disorder, via the SCID
* diagnosed with current Substance Use Disorder, via the SCID
* pose an imminent risk of self-harm or harm to others, assessed via the C-SSRS
* exhibit behavioral disturbance (e.g., aggression, mild-moderate cognitive impairment) that would significantly interfere with study participation, assessed by clinical research personnel

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Average self-reported working alliance measured by Working Alliance Inventory (WAI) | Weeks 1-8 CBT+ visits
  Working Alliance Inventory-Short Revised (WAI) is a 12-item survey on experiences over a therapy session and connection with a therapist. It consists of three subscales: tasks, goals, and therapist-client bond. The Goal, Task, and Bond domains each have scores ranging from 5 to 20. Higher scores indicate a better therapeutic alliance.
Average change in self-reported behavioral activation measured by Behavioral Activation for Depression Scale (BADS) | Intake, Weeks 1-8 CBT+ visits, final, 12-week follow up, 1-year follow-up
  The Behavioral Activation for Depression Scale (BADS) will be used to assess changes in behavioral activity. The scale is designed to be administered weekly to measure changes over the course of Behavioral Activation for depression. It consists of 25 questions that inquire about Activation, Avoidance/Rumination, Work/School Impairment, and Social Impairment (sub-scaled). A total score (all subscales summed) will be used as a primary outcome in this study.

SECONDARY OUTCOMES:
Changes in clinician-rated depression symptoms measured by GRID-Hamilton Depression Rating Scale (GRID-HAM-D) | Intake, final, 12-week follow up, 1-year follow up
  The GRID-HAM-D is a clinician-completed questionnaire that will be used to rate depressive symptom severity. The questionnaire is designed for adults and is used to rate the intensity and frequency of depressive symptoms by probing mood, feelings of guilt, suicidal ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. As recommended by the Depression Rating Scale Standardization Team, Clinical Interviewers will follow the Structured Interview Guide and use GRID scoring, in which dimensions of intensity and frequency of a symptom are rated independently for each item. Higher scores reflect greater symptom severity, categorized as Normal (0-7), Mild Depression (8-13), Moderate Depression (14-18), Severe Depression (19-22), and Very Severe Depression (>23).
Change in self-reported depression symptoms measured by Patient Health Questionnaire-9 (PHQ-9) | Intake, weeks 1-8 CBT+ visits, final, 12-week follow up, 1-year follow-up
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-question self-report instrument used to assess presence and severity of depressive symptoms, with scores categorized 0-4, 5-9, 10-14, 15-19, and 20-27 as minimal, mild, moderate, moderately severe, and severe depression, respectively.
Change in MDD diagnosis measured by Structured Clinical Interview for DSM-5 Disorders (SCID) | Intake, final, 12-week follow up, 1-year follow up
  The SCID is a clinician-administered semi-structured interview guide for making diagnoses according to the diagnostic criteria published in the American Psychiatric Association's Diagnostic and Statistical Manual for Mental Disorders (DSM-5). It provides diagnoses for depressive and bipolar disorders, schizophrenia spectrum and other psychotic disorders, substance use disorders, anxiety disorders (panic disorder, agoraphobia, social anxiety disorder, generalized anxiety disorder),obsessive-compulsive disorder, posttraumatic stress disorder, attention-deficit/hyperactivity disorder, and adjustment disorder.
Change in suicidal thoughts measured by the Columbia-Suicide Severity Rating Scale (CSSRS) | Intake, weeks 1-8 CBT+ visits, final, 12-week follow up, 1-year follow-up
  The C-SSRS will be used to assess and monitor suicide ideation and behavior. The severity of the ideation subscale is rated on a 5-point ordinal scale: 1 = wish to be dead, 2 = nonspecific active suicidal thoughts, 3 = suicidal thoughts with methods, 4 =suicidal intent, and 5 = suicidal intent with plan. Suicide behaviors are rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and non-suicidal,self-injurious behavior.
Average anhedonia measured by Dimensional Anhedonia Rating Scale (DARS) | Weeks 1-8 CBT+ visits (repeated 3 times [before exercise/calm condition, immediately after exercise/calm condition, and after therapy]), final, 12-week follow up, 1-year follow up
  The DARS is a self-report measure that assesses state anhedonia across multiple domains. DARS is a 17-item survey on state anhedonia divided into four domains: hobbies, food/drink, social activities, and sensory experiences. Subjects must list two activities within each of these categories that they consider their favorite and then respond to questions regarding their interest in/enjoyment of those activities on a 5-point Likert scale from "Not at all" to "Very much." During pre/post-administration, participants will be asked to respond to how they are feeling "right now."
Average anhedonia measured by an Anhedonia Visual Analogue Scale (Anhedonia VAS) | Weeks 1-8 CBT+ visits (repeated 3 times [before exercise/calm condition, immediately after exercise/calm condition, and after therapy]), final, 12-week follow up, 1-year follow up
  An anhedonia Visual Analog Scale [VAS] with 0 indicating 'No pleasure at all' and 100 indicating 'Greatest pleasure imaginable' will be used to measure anhedonia. In past research by the PI, correlations between the DARS and VAS were 0.49-0.69 indicating a moderate-to-strong agreement between the measures. The VAS will be used to provide a supplementary assessment of anhedonia.
Serum brain derived neurotrophic factor (BDNF) | Weeks 1, 4, and 8 CBT+ visits (before exercise/calm condition, immediately after exercise/calm condition, and after therapy)
  Serum BDNF will be quantified from a standard blood draw. Blood samples collected during Visits 1, 4, and 8 will be allowed to clot for 30 minutes and then centrifuged for ten minutes at 5500 RPM and 4 ◦C. Following centrifugation, blood serum will be extracted with samples stored at -80 ◦C until BDNF analysis. Enzyme-linked immunosorbent assay (ELISA) kits will measure the concentration of total BDNF in the serum according to the manufacturer's instructions. Each blood sample will be run in duplicate and averaged.
Change in monitor-assessed physical activity measured by accelerometry | Intake, weeks 4 & 8 CBT+ visits (monitors worn 1 week following each time point)
  Participants will place an activPAL on the midline of the thigh on either leg and wear the monitor during all waking hours, removing it only for water-based activities (e.g., swimming). For data to be valid, the monitor must have been worn for 20 hours on at least 4 days, including a minimum of 3 weekdays and 1 weekend day. Sleep time will be parsed out from each day's sitting/lying time automatically using PALanalysis. From these data, average minutes of sitting per day will be used to assess total sedentary time, minutes of stepping time with a cadence ≥75 and <100 will be used to assess minutes of light-intensity physical activity and minutes of stepping time with a cadence ≥100 will be used to assess minutes of moderate to vigorous physical activity (MVPA).
Change in self-reported physical activity measured by the International Physical Activity Questionnaire - Short Form (IPAQ-SF) | Intake, week 4 CBT+ visit, final, 12-week follow up, 1-year follow up
  The IPAQ is a physical activity questionnaire that inquires about average amounts of walking, moderate physical activity, vigorous physical activity, and sitting time per week.
Change in quality of life measured by the 36-Item Short Form Health Survey (SF-36) | Intake, week 4 CBT+ visit, final, 12-week follow up, 1-year follow up
  The SF-36 assesses health-related quality of life. It consists of eight scaled scores (including vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The higher the score the less disability (i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability).
Change in anxiety measured by Generalized Anxiety Disorder 7 (GAD-7) | Intake, week 4 CBT+ visit, final, 12-week follow up, 1-year follow up
  Generalized Anxiety Disorder 7 (GAD-7) is a self-reported questionnaire for measuring generalized anxiety disorder. GAD-7 has seven items, which measure the severity of various signs of GAD according to reported response categories of: Not at all (0 points), Several days (1 point), More than half the days (2 points), and Nearly every day (3 points), with scores of 5, 10, and 15 as cut-off points for mild, moderate and severe anxiety, respectively.
Average automatic thoughts measured by Automatic Thoughts Questionnaire (ATQ) | Intake, weeks 1-8 CBT+ visits, final, 12-week follow up, 1-year follow-up
  The ATQ is a 30-item instrument that measures the frequency of automatic negative statements about the self. Each item is rated on the frequency of an occurrence from "not at all" to "all the time". Total scores are the sum of all 30 items, with higher totals indicating a higher level of automatic negative self-statements.
Average session effectiveness measured by Session Evaluation Questionnaire (SEQ) | Weeks 1-8 CBT+ visits
  Session Evaluation Questionnaire (SEQ) will be used to evaluate session effectiveness. This includes responses to twenty-one items in a 7-point bipolar adjective format questionnaire to assess how the client feels about each CBT session. The questionnaire assesses session depth, smoothness, positivity, and arousal. An overall score of the average of the values across each subscale will be used in this study.
Average Lyssn generated scores | Weeks 1-8 CBT+ visits
  Lyssn is an AI-powered assessment platform for recording and managing session files, and all clinical interviews and therapy sessions will be recorded on the Lyssn platform. Lyssn will process the audio files from therapy sessions to generate session-level data regarding collaboration and empathy as metrics related to the primary client ratings of working alliance, as well as generating CTRS fidelity metrics which will be used in the ongoing supervision and fidelity monitoring of all sessions.
Nature Connectedness Index (NCI) | Intake, Weeks 1, 4, and 8 CBT+ visits (before exercise/calm condition, immediately after exercise/calm condition, and after therapy)
  The NCI consist of 6 questions pertaining to nature connectedness. Participants respond using a 7-point Likert scale, ranging from 1 (Strongly Disagree) to 7 (Strongly Agree), with higher scores indicating greater levels of nature connectedness.

OTHER OUTCOMES:
Health History Questions | Intake
  Health history will be self-reported. In addition, participants will be asked to list their current medications.
Demographic Questionnaire | Intake
  Demographic characteristics including age, sex, race, education, marital status, occupational status, and household income will be recorded or measured to characterize the sample.
Adverse Childhood Experience Survey (ACES) | Intake
  The ACES consists of 16 questions pertaining to the respondents' first 18 years of life. Participants respond with yes or no regarding if a childhood adverse event occurred. Adverse events questions are grouped by categories. Participants are scored for each event category they are exposed to with scores ranging from 0 (unexposed) to 7 (exposed to all categories).

CONTACTS AND LOCATIONS:
Locations (1):
- Iowa State University, Ames, Iowa, United States

REFERENCES:
- [Derived] Meyer JD, Kelly SJE, Gidley JM, Lansing JE, Smith SL, Churchill SL, Thomas EBK, Goldberg SB, Abercrombie HC, Murray TA, Wade NG. Protocol for a randomized controlled trial: exercise-priming of CBT for depression (the CBT+ trial). Trials. 2024 Oct 7;25(1):663. doi: 10.1186/s13063-024-08495-x. PMID 39375728

DOCUMENTS (1):
  • Informed Consent Form (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT06001346/ICF_000.pdf